CLINICAL TRIAL: NCT02885129
Title: Development of the General Scale Observance for Chronic Diseases (EGOMAC)
Brief Title: Development of the General Scale Observance for Chronic Diseases
Acronym: EGOMAC
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Other Study IDs: PSS 2014/EGOMAC-GUILLEMIN/SR
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Chronic Diseases
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective is to assess the measurement characteristics (validity, reproducibility) and the invariance of EGOMAC scale in a population of consultants in diabetology, cardiology and rheumatology hospital and liberal and hospital oncology and Infectious disease, by following the evolution of patient compliance at D0 and D15.

The second objective is to assess the sensitivity to change of scale EGOMAC following developments compliance 3 months.

DETAILED DESCRIPTION:
During a routine appointment (D0), the patient filled a newsletter and a questionnaire to complete.

The doctor collects medical informations for the case report form.

At the end of the first consultation (D0), an additional EGOMAC scale and a stamped envelope is delivered to the patient by asking him to fill that scale to 15 days and return it by Post Office (reproducibility study).

Finally, a new scale will be addressed to the patient at the end of 3 months, which will return by Post Office too (stability study).

ELIGIBILITY:
Inclusion Criteria:

* patient age of 18 years
* from routine patient counseling
* with at least one of these diseases : heart failure, hypertension, coronary disease, type 2 diabetes, osteoarthritis of the knee or hip, osteoporosis, inflammatory rheumatism (rheumatoid arthritis, spondyloarthropathy), cancer ( with only non-hormonal oral anti cancer treatments) and HIV.
* patient can read the French language in order to complete the self -administered questionnaire
* patient agreeing to participate in the study

Exclusion Criteria:

* patient treated for more than 3 conditions mentioned in the inclusion criteria (
* patient receiving no drug prescription or recommendation of lifestyle or diet (for example consultationpurely diagnostic ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of consultants in diabetology, cardiology and rheumatology hospital and liberal and hospital oncology and Infectious disease
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2014-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
EGOMAC questionnaire | baseline
Change in EGOMAC questionnaire | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Francis GUILLEMIN, MD, PhD, Principal Investigator — CHRU Nancy
Locations (1):
- Central hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
open to partnership